CLINICAL TRIAL: NCT06442345
Title: Real-time Pneumocystis Jirovecii Genotyping to Support Clinical Decision Making in the Management of Nosocomial Outbreaks
Brief Title: Pneumocystis Jirovecii Genotyping
Status: Not yet recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23PA004
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pneumocystis Pneumonia
Keywords: PCP; Genotyping
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We share our lives with microorganisms, and these generally do not pose a problem if an individual is healthy with a normal immune system. However, if the immune system was not functioning properly (e.g., cancer patients), they are at risk of infection. One microorganism, a fungus called Pneumocystis jirovecii (PCP), can cause severe chest infections in patients without properly functioning immune systems, leading to hospitalisation and death if untreated. If patients remain without a functioning immune system, they have a greater chance of repeated infection.

PCP spreads through air from person-to-person and can survive on environmental surfaces. Patients can be infected after contact with these surfaces. Hospitals have a responsibility to ensure PCP infected patients do not pass it on to other unwell patients. In cases where PCP has infected multiple patients, knowing if the same fungi has been passed along (or transmitted) from patient-to-patient is vital in understanding if there is an outbreak in the hospital. Understanding how similar (the relatedness) the PCP strain is allows healthcare workers to detect any transmission between patients or the environment.

To understand how related each patient's PCP infection is we will utilise a laboratory test called multilocus sequence typing (MLST). This test looks at sections of the fungi's genetic code using deoxyribonucleic acid (DNA) sequencing to create a code (genotype) which tells us how related one PCP is to others tested, allowing comparison between patients and ultimately spotting transmission.

Our aim is to develop this sequencing test using PCP positive patient samples and ensure it performs to high-quality standards. Surplus material from seventy known PCP positive patient samples will be tested. Each sample will be analysed to see if the DNA genotype matches or is similar to other patient samples we have tested, helping to understand how PCP may spread between patients.

DETAILED DESCRIPTION:
We share our lives with microorganisms, and these generally do not pose a problem if an individual is healthy with a normal immune system. However, if the immune system was not functioning properly (e.g., cancer patients), they are at risk of infection. One microorganism, a fungus called Pneumocystis jirovecii (PCP), can cause severe chest infections in patients without properly functioning immune systems, leading to hospitalisation and death if untreated. If patients remain without a functioning immune system, they have a greater chance of repeated infection.

PCP spreads through air from person-to-person and can survive on environmental surfaces. Patients can be infected after contact with these surfaces. Hospitals have a responsibility to ensure PCP infected patients do not pass it on to other unwell patients. In cases where PCP has infected multiple patients, knowing if the same fungi has been passed along (or transmitted) from patient-to-patient is vital in understanding if there is an outbreak in the hospital. Understanding how similar (the relatedness) the PCP strain is allows healthcare workers to detect any transmission between patients or the environment.

To understand how related each patient's PCP infection is we will utilise a laboratory test called multilocus sequence typing (MLST). This test looks at sections of the fungi's genetic code using deoxyribonucleic acid (DNA) sequencing to create a code (genotype) which tells us how related one PCP is to others tested, allowing comparison between patients and ultimately spotting transmission.

Our aim is to develop this sequencing test using PCP positive patient samples and ensure it performs to high-quality standards. Surplus material from seventy known PCP positive patient samples will be tested. Each sample will be analysed to see if the DNA genotype matches or is similar to other patient samples we have tested, helping to understand how PCP may spread between patients.

ELIGIBILITY:
Inclusion Criteria:

* Total nucleic acid extracts from adult patients (over 18 years old) with a positive PCP diagnosis (& detected at > 50 copies/10ul) from routine respiratory panel testing.

Exclusion Criteria:

* Total nucleic acid extracts from patients with a negative PCP diagnosis from routine respiratory panel testing
* Total nucleic acid extracts from non-adult patients (under 18 years old).
* PCP positive total nucleic extract samples with < 50 copies/10ul.
* Patients included on the UK National Opt-Out register

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults PCP positive patients over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Objective 1: Development of a MLST PCP genotyping assay within NUH. | 18 months
  The previously published MLST scheme by Pasic et al (2020) using alleles β-TUB, CYB, mt26S and SOD will be assessed, with each allele optimised and verified for implementation for Objective 2.

SECONDARY OUTCOMES:
Objective 2: Analyse PCP positive patient samples and identify the PCP genotype, assessing links between patient metadata and genotype | 18 months
  Following successful implementation of the MLST assay, up to 70 known PCP positive total nucleic acid samples will be tested using the MLST assay. Genotypes will be identified and phylogenetic analysis performed to assess the relatedness of the population. From this we will assess for possible transmission events between patients using patient metadata and hospital bed movements/clinic visits. Furthermore, data analysis will help understand if certain PCP genotypes are more likely to occur in specific patient groups, and if there are links to disease severity, mortality & transmission.